CLINICAL TRIAL: NCT02019849
Title: Post Market Clinical Follow-Up of Plasmafit® Cup
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1213
Record Dates: First submitted 2013-12-04; First posted 2013-12-24 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Total Hip Arthroplasty
Keywords: THA, Plasmafit®

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Plasmafit® Total Hip Arthroplasty
  Interventions: Device: Plasmafit® Total Hip Arthroplasty

INTERVENTIONS:
Device: Plasmafit® Total Hip Arthroplasty

SUMMARY:
Twelve months follow-up of implant survival and clinical and radiological follow-up of Plasmafit® Cup.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age 18 years
* Indication for cementless total hip arthroplasty
* Patient consent for study participation
* Physical and mental willingness to participate at clinical and radiological follow-up

Exclusion Criteria:

* Patient not available for follow-up
* Increased anesthetics risks according to the "American Society of Anesthesiology": ASA IV
* Tumor
* Alcohol or drug abuse
* Permanent cortisone therapy
* Clinically relevant infection
* Pregnancy or planned pregnancy
* Prior interventions like osteotomy, fracture treatment or prior THA at the concerned hip
* Acute fracture at the concerned hip
* Patients needing a cemented hip arthroplasty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Specialist Clinical Centre
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-06-18 (Actual); Primary Completion 2012-10-04 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
Implant Survival Rates | 10 years
  Implant survival is analysed at follow-up examinations at 3 months, 12 months, 5 years and 10 years

SECONDARY OUTCOMES:
Osteolysis | 3 months, 12 months, 5 years, 10 years
  Radiological Outcome
Ossifications | 3 months, 12 months, 5 years, 10 years
  Radiological Outcome
Implant Position | 3 months, 12 months, 5 years, 10 years
  Radiological Outcome
Migration of Plasmafit® | 3 months, 12 months, 5 years, 10 years
  Radiological Outcome
Clinical Outcome | 3 months, 12 months, 5 years, 10 years
  Harris Hip Score

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Vulpius-Klinik Bad Rappenau, Bad Rappenau
  - Diakonie-Klinikum Stuttgart, Stuttgart